CLINICAL TRIAL: NCT04414033
Title: Bubble: A New VR-AI Way of Treatment for Hot Flashes in Women With Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bar-Ilan University, Israel (Other)
Collaborators: Hematology and Oncology Specialists (Other)
Responsible Party: Principal Investigator, Danny Horesh, Senior lecturer and head of the Trauma and Stress Research Lab at Bar-Ilan University's Department of Psychology, Bar-Ilan University, Israel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22012020
Record Dates: First submitted 2020-05-15; First posted 2020-06-04 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Hot Flashes; Breast Cancer
MeSH Terms: conditions — Hot Flashes; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- research group (Experimental)
  Interventions: Device: Bubble: A New VR-AI Way of Treatment for Hot Flashes

INTERVENTIONS:
Device: Bubble: A New VR-AI Way of Treatment for Hot Flashes — Bubble Bubble is a virtual reality (VR) mobile application. Bubble offers a psychological intervention based upon cognitive behavioral therapy (CBT) and mindfulness-based stress reduction (MBSR) protocols. The bubble mobile application offers the intervention in a virtual reality (VR) coaching environment and in a winter wonderland setting called Frosty. Frosty provides both a virtual reality winter wonderland experience as well as guided meditation. The cold, winter-like experience is designed to help patients calm down and feel cooler.

SUMMARY:
This study evaluates the potential of a unique artificial intelligence-virtual reality intervention called Bubble, to reduce the number and intensity of hot flashes and their accompanying psychological symptoms in women, aged 28-55, with breast cancer. A sample of 37 women with breast cancer were selected to the study. Participants were asked to answer a survey before and after using Bubble. The treatment period was 24 days. The findings are positive and show that the use of Bubble help to reduce several psychological symptoms connected to hot flashes.

DETAILED DESCRIPTION:
Breast cancer is the most common cancer in women and the leading cause of death in women aged < 55 years . Hot flashes are experienced by about 52% of perimenopausal women. After breast cancer, this may increase to 70%. Hot flash is a subjective sensation of heat that is associated with objective signs of cutaneous vasodilatation and a subsequent drop in core temperature. The hot flash may be accompanied by physiological symptoms as sweating, flashing, palpitations, and night sweat. As well as by psychological symptoms as anxiety, irritability, and even panic. Hot flashes and night sweats (HF/NS) affect 65-85% of breast cancer survivors and are associated with sleep problems and reduced quality of life.

It is well known that estrogen largely alleviates vasomotor symptoms, however concerns regarding its use in women, with or without breast cancer, has led to extensive research efforts to find well tolerated and efficient nonhormonal interventions. Postmenopausal women and breast cancer survivors experience psychological, spiritual, sleep, and cognitive dysfunction beyond what could be attributable to vasomotor symptoms alone. Therefore, an integrative intervention that can address multiple symptoms is an important patient-centric strategy.

These days a growing body of research has been dedicated to mind-body interventions. These interventions include yoga, hypnosis, relaxation-training/paced respiration, mindfulness-based stress reduction (MBSR), and cognitive behavioral therapy (CBT). In practice, a previous study demonstrated that distressing or problematic hot flashes were predicted by depression, anxiety, and low self-image, but not by the frequency of the hot flashes. Therefore, women with the same amount of hot flashes may have different and diverse emotional responses to their hot flashes. This psychosocial aspect plays a role in the distress or can be related to the symptom as well as to the person's will to do something about his situation. Cognitive behavioral therapy has a long and well documented history of efficacy related to distress, sleep, and psychological aspects of coping with many of life's challenges. A study showed that a brief, mindfulness-based intervention demonstrated preliminary short-term efficacy in reducing stress, behavioral symptoms, and proinflammatory signaling in younger breast cancer survivors. Also, research indicated that relaxation training reduced the incidence and severity of hot flashes and the distress caused by the flashes in women with primary breast cancer compered to control group.

Virtual reality (VR) is a computer technology that uses virtual reality headsets or multi-projected environments, sometimes in combination with physical environments or props, to generate realistic images, sounds and other sensations that simulate a user's physical presence in a virtual or imaginary environment. Today there are two main categories of VR, immersive and non-immersive. Immersion or presence can be regarded as a variable that can influence the effects on the attention of users. Full immersion is reached by a head mounted display, which blocks the users' view of the real world and presents patients with a view of a computer-generated world instead. This technology may offer subjects a safe environment.

A review of 19 studies reporting the use of VR in therapies related to cancer patients showed that four out of eight studies that evaluated bio-physiological outcomes found significant differences in pulse rate, showing lower heart rate in the VR group compared with the non-treatment control group. Furthermore, all studies evaluating the efficacy of VR on different psychological variables found a significant improvement following treatment. In addition, there have been studies of virtual reality in women receiving chemotherapy, older women with breast cancer receiving chemotherapy, adults with breast, colon and lung cancer receiving chemotherapy, and older children receiving chemotherapy. Results of these interventions have been positive, with patients reporting to decreased psychological distress, perception that treatment times were shortened and a belief that treatment with virtual reality was better than chemotherapy alone. Importantly, patients generally did not report cyber sickness (i.e., nausea and discomfort that can last for hours after participating in VR applications) and the VR intervention was easy to implement.

Previous findings in the field of body-mind treatments, and specifically VR as a treatment for women with breast cancer, have led to the current study, which aimed to evaluate the Bubble, a new VR-AI way of treatment specifically tailored for improving symptoms associated with hot flashes in female cancer patients. As previous findings in the field showed the advantages of VR, CBT and mindfulness as treatments for women with cancer or for women who suffer from hot flashes, they are not specific to hot flashes caused by cancer nor not combining the three methods together. In this study we are trying to understand the effect of CBT and mindfulness treatment when given with a VR technology. Specifically, we tried to explore the effect of this combined type of treatment on women who suffer from hot flashes caused by cancer. Furthermore, the current study tries to understand what method work for whom and hence we recruited younger and older women and didn't focused only on one age group.

This pilot study evaluated the potential of a unique artificial intelligence-virtual reality intervention called Bubble, to reduce the number and intensity of hot flashes and their accompanying psychological symptoms in women, aged 28-55, with breast cancer. A repeated measures design was used to answer the following questions: (1) Is AI-VR an effective intervention for reducing hot flashes in women with breast cancer? (2) Is AI-VR intervention decreases the intensity and/or frequency of symptoms associated with hot flashes in women with breast cancer?

Based on past research, as well as our own pilot data collected from focus groups (detailed in the procedure section), we hypothesized that the use of Bubble will lead to an improvement decrease intensity of hot flashes and the psychological symptoms connecting to them (stress, psychopathology level), as well as improve life and sleep quality.

ELIGIBILITY:
Inclusion Criteria:

* Females between the ages of 18 and 60
* Having an existing diagnosis of breast or ovarian cancer
* Receiving standard-of-care chemotherapy, endocrine therapy or estrogen blocking anti-cancer treatment
* The woman reported experiencing hot flashes at least once per day for a duration of at least 7 days prior to the beginning of the study and hot flashes for at least 30 days prior to the beginning of the study
* No chronic migraine headaches, seizure disorders, serious vestibular disorders, or pathological vertigo
* No serious psychiatric disorders
* Not pregnant
* No current substance abuse
* Not participating in other forms of therapy
* Not using medical marijuana.

Exclusion Criteria:

* women aged 28-55 with breast cancer suffering from hot flashes

Ages: 28 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Demographic and background (disease & treatment-elated) information | Through study completion, an average of 1 month
  A form was used to assess demographic information, including birth date, race, education, marital status, employment status, and household income. Women also were asked to record their height and weight, which was used to calculate body mass index. Routine information regarding date of diagnosis, stage of disease, and types and dates of cancer treatments was obtained from medical records
HFRDIS, The Hot Flash Related Daily Interference Scale | Through study completion, an average of 1 month, before the manipulation
  The Hot Flash Related Daily Interference Scale (HFRDIS;Carpenter, 2001) is a 10-item scale measuring the degree to which hot flashes interfere with nine daily activities; the tenth item measures the degree hot flashes interfere with overall quality of life. The HFRDIS was developed to include daily life activities specific to the impact of hot flashes. Participants rate the degree to which hot flashes have interfered with each item during the previous week using a 0 (do not interfere) to 10 (completely interfere) point scale. A total score is computed by summing items. Higher scores indicate higher interference due to hot flashes and thus, greater impact on quality of life.
HFRDIS, The Hot Flash Related Daily Interference Scale | Through study completion, an average of 1 month, after the manipulation
  The Hot Flash Related Daily Interference Scale (HFRDIS;Carpenter, 2001) is a 10-item scale measuring the degree to which hot flashes interfere with nine daily activities; the tenth item measures the degree hot flashes interfere with overall quality of life. The HFRDIS was developed to include daily life activities specific to the impact of hot flashes. Participants rate the degree to which hot flashes have interfered with each item during the previous week using a 0 (do not interfere) to 10 (completely interfere) point scale. A total score is computed by summing items. Higher scores indicate higher interference due to hot flashes and thus, greater impact on quality of life.
HFRS, The Hot Flash Rating Scale | Through study completion, an average of 1 month, before the manipulation
  measures the frequency and intensity of hot flashes and night sweats per day and per week. It also estimates chronicity and average duration of the hot flashes, as well as provides rating on three separate ten-point scales (1/10 being the least and 10/10 being the most) for the amount of distress, the extent to which HFs interfered with daily life and the degree to which HFs were a problem in patients' lives. A higher score indicates more HF per day.
HFRS, The Hot Flash Rating Scale | Through study completion, an average of 1 month, after the manipulation
  measures the frequency and intensity of hot flashes and night sweats per day and per week. It also estimates chronicity and average duration of the hot flashes, as well as provides rating on three separate ten-point scales (1/10 being the least and 10/10 being the most) for the amount of distress, the extent to which HFs interfered with daily life and the degree to which HFs were a problem in patients' lives. A higher score indicates more HF per day.
PSS, The Perceived Stress Scale | Through study completion, an average of 1 month, before the manipulation
  a self-reported questionnaire that was designed to measure the degree to which situations in one's life over the past week are appraised as unpredictable, uncontrollable and overwhelming. It posits that people appraise potentially-threatening or challenging events in relation to their available coping resources. Items are rated on a Likert scale ranging from 0 (never) to 4 (very often). A higher score indicates a greater degree of perceived stress.
PSS, The Perceived Stress Scale | Through study completion, an average of 1 month, after the manipulation
  a self-reported questionnaire that was designed to measure the degree to which situations in one's life over the past week are appraised as unpredictable, uncontrollable and overwhelming. It posits that people appraise potentially-threatening or challenging events in relation to their available coping resources. Items are rated on a Likert scale ranging from 0 (never) to 4 (very often). A higher score indicates a greater degree of perceived stress.
K10, The Kessler Psychological Distress Scale | Through study completion, an average of 1 month, before the manipulation
  10-item measure of psychological distress in the past month, which reliably predicts the presence of a current depressive or anxiety disorder at a cut-off score of 17. The K10 is a 10-item questionnaire rated on a five-point Likert-type scale (from "none of the time" = 1 to "all of the time" = 5). A higher score indicates a greater degree of distress.
K10, The Kessler Psychological Distress Scale | Through study completion, an average of 1 month, after the manipulation
  10-item measure of psychological distress in the past month, which reliably predicts the presence of a current depressive or anxiety disorder at a cut-off score of 17. The K10 is a 10-item questionnaire rated on a five-point Likert-type scale (from "none of the time" = 1 to "all of the time" = 5). A higher score indicates a greater degree of distress.
B-IPQ, The Brief Illness Perception Questionnaire | Through study completion, an average of 1 month, before the manipulation
  is designed to provide simple and rapid assessment of illness perceptions, using single items on a scale from 1-10 to assess each item including; perceived consequences, timeline (acute vs chronic), amount of perceived personal control, treatment control, identity (symptoms), concern about the illness, coherence of the illness and emotional representation of the illness.
B-IPQ, The Brief Illness Perception Questionnaire | Through study completion, an average of 1 month, after the manipulation
  is designed to provide simple and rapid assessment of illness perceptions, using single items on a scale from 1-10 to assess each item including; perceived consequences, timeline (acute vs chronic), amount of perceived personal control, treatment control, identity (symptoms), concern about the illness, coherence of the illness and emotional representation of the illness.
PSQI, The Pittsburgh Sleep Quality Index | Through study completion, an average of 1 month, before the manipulation
  a retrospective self-report questionnaire that measures sleep quality over the previous month. Seven clinically derived domains of sleep difficulties (sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medications, and daytime dysfunction) are assessed. The PSQI global score allowed discriminating between healthy controls and patients, and between groups of patients affected by different pathologies. Results also indicated that the best cut-off score (differentiating "good" from "bad" sleepers) is 5.
PSQI, The Pittsburgh Sleep Quality Index | Through study completion, an average of 1 month, after the manipulation
  a retrospective self-report questionnaire that measures sleep quality over the previous month. Seven clinically derived domains of sleep difficulties (sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medications, and daytime dysfunction) are assessed. The PSQI global score allowed discriminating between healthy controls and patients, and between groups of patients affected by different pathologies. Results also indicated that the best cut-off score (differentiating "good" from "bad" sleepers) is 5.
WHOQOL-BREF, The World Health Organization Quality of Life Scale | Through study completion, an average of 1 month, before the manipulation
  assesses individuals' perception of their position in life in the context of the culture and value systems in which they live and in relation to their goals, expectations, standards and concerns. The WHOQOL-BREF is a 26-item version of the WHOQOL-100 scale, and as the WHOQOL-100 it includes four domains: physical, psychological, social and environmental QOL and 5-point response scales (5,Very satisfied-1,Very dissatisfied;1,Not at all-5,Extremely; 1,Not at all-5,Completely; and 1,Never-5,Always) and Domain scores are scaled in a positive direction (i.e. higher scores denote higher quality of life).
WHOQOL-BREF, The World Health Organization Quality of Life Scale | Through study completion, an average of 1 month, after the manipulation
  assesses individuals' perception of their position in life in the context of the culture and value systems in which they live and in relation to their goals, expectations, standards and concerns. The WHOQOL-BREF is a 26-item version of the WHOQOL-100 scale, and as the WHOQOL-100 it includes four domains: physical, psychological, social and environmental QOL and 5-point response scales (5,Very satisfied-1,Very dissatisfied;1,Not at all-5,Extremely; 1,Not at all-5,Completely; and 1,Never-5,Always) and Domain scores are scaled in a positive direction (i.e. higher scores denote higher quality of life).

CONTACTS AND LOCATIONS:
Locations (1):
- Bar Ilan University, Ramat Gan, Israel

REFERENCES:
- See also: Andrews, G., & Slade, T. (2001). Interpreting scores on the Kessler Psychological Distress Scale (K10). Australian and New Zealand Journal of Public Health, 25(6), 494-497. — https://doi.org/10.1111/j.1467-842X.2001.tb00310.x
- See also: Blumel, J. E., Castelo-Branco, C., Binfa, L., Gramegna, G., Tacla, X., Aracena, B., … Sanjuan, A. (2000). Quality of life after the menopause: A population study. Maturitas, 34(1), 17-23. — https://doi.org/10.1016/S0378-5122(99)00081-X
- See also: Buysse, D. J., Reynolds, C. F., Monk, T. H., Berman, S. R., & Kupfer, D. J. (1989). The Pittsburgh sleep quality index: A new instrument for psychiatric practice and research. Psychiatry Research, 28(2), 193-213 — https://doi.org/10.1016/0165-1781(89)90047-4
- See also: Fenlon, D. R., Corner, J. L., & Haviland, J. S. (2008). A Randomized Controlled Trial of Relaxation Training to Reduce Hot Flashes in Women with Primary Breast Cancer. Journal of Pain and Symptom Management, 35(4), 397-405 — https://doi.org/10.1016/j.jpainsymman.2007.05.014
- See also: Hardy, C. (2017). The Hot Flash Related Daily Interference Scale: Cutoffs, minimally important differences, and a revised short version. Menopause, 24(8), 869-870. — https://doi.org/10.1097/GME.0000000000000933
- See also: Kadakia, K. C., Loprinzi, C. L., & Barton, D. L. (2012). Hot flashes: The ongoing search for effective interventions. Menopause: The Journal of The North American Menopause Society, 19(7), 719-721. — https://doi.org/10.1097/gme.0b013e3182578d31
- See also: Lee, E.-H. (2012). Review of the Psychometric Evidence of the Perceived Stress Scale. Asian Nursing Research, 6(4), 121-127. — https://doi.org/10.1016/j.anr.2012.08.004
- See also: Nilsson, S., Finnström, B., Kokinsky, E., & Enskär, K. (2009). The use of Virtual Reality for needle-related procedural pain and distress in children and adolescents in a paediatric oncology unit. European Journal of Oncology Nursing, 13(2), 102-109 — https://doi.org/10.1016/j.ejon.2009.01.003
- See also: Schneider, Susan M., & Hood, L. E. (2007). Virtual Reality: A Distraction Intervention for Chemotherapy. Oncology Nursing Forum, 34(1), 39-46 — https://doi.org/10.1188/07.ONF.39-46
- See also: Schneider, Susan M., Prince-Paul, M., JoAllen, M., Silverman, P., & Talaba, D. (2004). Virtual Reality as a Distraction Intervention for Women Receiving Chemotherapy. Oncology Nursing Forum, 31(1), 81-88. — https://doi.org/10.1188/04.ONF.81-88
- See also: Skevington, S. M., Lotfy, M., & O'Connell, K. A. (2004). The World Health Organization's WHOQOL-BREF quality of life assessment: Psychometric properties and results of the international field trial. — https://doi.org/10.1023/B:QURE.0000018486.91360.00
- See also: Stearns, V., Ullmer, L., Lopez, J. F., Smith, Y., Isaacs, C., & Hayes, D. F. (2002). Hot flushes. The Lancet, 360(9348), 1851-1861 — https://doi.org/10.1016/S0140-6736(02)11774-0
- See also: Tatrow, K., & Montgomery, G. H. (2006). Cognitive Behavioral Therapy Techniques for Distress and Pain in Breast Cancer Patients: A Meta-Analysis. Journal of Behavioral Medicine, 29(1), 17-27 — https://doi.org/10.1007/s10865-005-9036-1
- See also: The World Health Organization quality of life assessment (WHOQOL): Position paper from the World Health Organization. (1995). Social Science & Medicine, 41(10), 1403-1409. — https://doi.org/10.1016/0277-9536(95)00112-K